CLINICAL TRIAL: NCT01641029
Title: Surveillance and Risk Factor Analysis of Community-Associated Uropathogen Antimicrobial Resistance Among Emergency Department Patients With Acute Pyelonephritis in the United States
Brief Title: Community-Associated Uropathogen Antimicrobial Resistance Among Emergency Department Patients With Acute Pyelonephritis
Status: Completed | Type: Observational
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 11H-770351
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Pyelonephritis
MeSH Terms: conditions — Pyelonephritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pyelonephritis: Patients > 18 years of age with flank pain and/or costovertebral angle tenderness, documented temperature in the emergency department of ≥38°C/100.4°F by any method of measurement, and clinically suspected acute pyelonephritis. Patients will be identified by their emergency department treating physicians.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention

SUMMARY:
Pyelonephritis is a serious infection that manifests with fever, back pain, nausea, and vomiting. In the U.S., it is estimated that there are 20 cases of pyelonephritis per 10,000 annually, with the highest incidence in young women. Escherichia coli (E. coli) causes over 80% of these infections. Over the last two decades, E. coli resistance has emerged to commonly prescribed antimicrobials, such as ampicillin and trimethoprim-sulfamethoxazole (TMP/SMX). Most recently, resistance to fluoroquinolones and strains producing extended-spectrum beta-lactamases (ESBL) have been observed. In order to better understand the evolution and current state of antibiotic resistance among E. coli urinary tract isolates so as to better inform treatment decisions, the investigators propose to conduct an investigation to: a) determine the prevalence of antimicrobial resistance among E. coli causing acute pyelonephritis in various patient groups, and specifically healthy community-dwellers with uncomplicated infections, b) determine the specific prevalence of fluoroquinolone-resistance and ESBL-producing E. coli, and c) determine potential risk factors for fluoroquinolone and ESBL-producing E. coli infections.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years of age with flank pain and/or costovertebral angle tenderness
* documented temperature in the emergency department of ≥38°C/100.4°F by any method of measurement,
* documented temperature in the emergency department of ≥38°C/100.4°F by any method of measurement,

Exclusion Criteria:

* complicated pyelonephritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from ten U.S. university-affiliated medical center emergency departments participating in a CDC-collaborative emerging infections sentinel network, EMERGEncy ID NET. Patients presenting with symptoms of acute uncomplicated pyelonephritis will be enrolled by treating physicians or study coordinators.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of antimicrobial resistant E. coli in the U.S. | July 2013-July 2014

CONTACTS AND LOCATIONS:
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States